CLINICAL TRIAL: NCT07308535
Title: EFFECTS OF TRAINING WITH STROBOSCOPIC GLASSES ON ATHLETIC PERFORMANCE IN VOLLEYBALL PLAYERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KA25/182
Record Dates: First submitted 2025-11-19; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Stroboscopic Visual Training; Physical Fitness
Keywords: Volleyball; stroboscopic glasses; athletic performance; physical fitness; visual training

STUDY DESIGN:
Intervention Model Description: In the study, individuals were evaluated face to face at the Turkish Volleyball Federation Beştepe Volleyball Hall. The evaluations lasted 30 minutes for each individual. After the sociodemographic information of the individuals in our study was recorded, individuals were divided into two groups as the experimental group and the control group using a computer numbering system. Necessary information and explanations were provided to individuals in the experimental group with Senaptec brand stroboscopic glasses (Beaverton, Oregon USA) before the application. Passing, reception and blocking training was performed with glasses in the stroboscopic glasses group. Training was performed without stroboscopic glasses in the control group. It was performed after the players' warm-up exercises for 3 sessions per week for 6 weeks. Since there was one stroboscopic glass, the evaluations were planned for 2 days, lasting 30 minutes for each individual. Reaction time, agility and anaerobic power were
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stroboscopic glasses group (Experimental): 27 volleyball players were evaluated at three times: pre-exercise, after 6 weeks and after 10 weeks regard to reaction time, agility, anaerobic performance, balance and coordination. Experimental group used stroboscopic glasses when doing exercise. Exercise program consisted lunge, jumping and balance exercises. Each exercise consisted 12 repetitions and 3 sets. Stroboscopic glasses were adjusted to 100 ms on/150 ms off flash level 3. This frequency are always preferred scientific research about stroboscopic visual training.
  Interventions: Device: stroboscopic visual training
- Control group (No Intervention): 27 volleyball players only exercised

INTERVENTIONS:
Device: stroboscopic visual training — 27 volleyball players were evaluated two times: pre-exercise and after 6 weeks. Reaction time, agility, anaerobic performance, balance and coordination were measured regard to athletic performance. Athletes using stroboscopic glasses perform exercise program. Exercise program consisted of lunge, balance and jumping exercises. Each exercise consisted of 12 repetitions and 3 sets. Stroboscopic glasses were adjusted to 100 ms on/150 ms off flash level 3. This frequency is always preferred in scientific research.
  Arms: stroboscopic glasses group

SUMMARY:
This study was conducted to investigate the effects of training with stroboscopic glasses on athletic performance in volleyball players. 54 male volleyball players participated in the study. Individuals were randomly divided into two groups as experimental group (n=27) and control group (n=27). Passing, reception and blocking exercises were performed paired with stroboscopic glasses in the experimental group and without glasses in the control group for 6 weeks. Measurements were made twice, before the exercise program and at the end of the 6-week exercise program. Reaction time was evaluated with the Human Benchmark test, agility with T agility test, anaerobic power with vertical jump, balance with Flamingo balance test, coordination with Hexagonal coordination test.

DETAILED DESCRIPTION:
In the study, individuals were evaluated face to face at the Turkish Volleyball Federation Beştepe Volleyball Hall. The evaluations lasted 30 minutes for each individual. After the sociodemographic information of the individuals in our study was recorded, individuals were divided into two groups as the experimental group and the control group using a computer numbering system. Necessary information and explanations were provided to individuals in the experimental group with Senaptec brand stroboscopic glasses (Beaverton, Oregon USA) before the application. Passing, reception and blocking training was performed with glasses in the stroboscopic glasses group. Training was performed without stroboscopic glasses in the control group. It was performed after the players' warm-up exercises for 3 sessions per week for 6 weeks. Since there was one stroboscopic glass, the evaluations were planned for 2 days, lasting 30 minutes for each individual. Reaction time, agility and anaerobic power were performed on the first day, and coordination and balance were performed on the second day. The evaluations were performed after the warm-up exercises. The evaluations were performed twice, before the training program and at the end of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male individuals between the ages of 18-35
* Being a professional volleyball player
* Not having undergone surgery in the last 6 months
* Not having any chronic, systemic or neuromuscular disease
* Not having any visual, cognitive or vestibular disorders

Exclusion Criteria:

* Individuals under the age of 18 and over the age of 35
* Female individuals
* Sedentary individuals
* Having visual, cognitive or vestibular disorders
* Having any chronic, systemic neuromuscular diseases

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Volleyball Players
Enrollment: 54 (Actual)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-05-11 (Actual); Study Completion 2025-05-24 (Actual)

PRIMARY OUTCOMES:
Reaction time | 6 weeks
  Human Benchmark Test
Agility | 6 weeks
  T Agility Test
Anaerobic Performance | 6 weeks
  Vertical Jumping
Balance | 6 weeks
  Flamingo Balance Test
Coordination | 6 weeks
  Hexagonal Coordination Test

CONTACTS AND LOCATIONS:
Overall Officials: Nihan Özünlü PEKYAVAŞ, PROFESSOR, Study Director — Baskent University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Research evaluated individual athletic performance. Volleyball team manager did not want to share individual performance data.

REFERENCES:
- [Result] Ramirez-Campillo R, Andrade DC, Nikolaidis PT, Moran J, Clemente FM, Chaabene H, Comfort P. Effects of Plyometric Jump Training on Vertical Jump Height of Volleyball Players: A Systematic Review with Meta-Analysis of Randomized-Controlled Trial. J Sports Sci Med. 2020 Aug 13;19(3):489-499. eCollection 2020 Sep. PMID 32874101
- [Result] Zwierko T, Tapia V, Vera J, Redondo B, Morenas-Aguilar MD, Garcia-Ramos A. Enhancing reactive agility in soccer: The impact of stroboscopic eyewear during warm-up across fatigued and non-fatigued conditions. Eur J Sport Sci. 2024 Dec;24(12):1798-1808. doi: 10.1002/ejsc.12224. Epub 2024 Nov 22. PMID 39578413
- [Result] Ahmadi M, Nobari H, Ramirez-Campillo R, Perez-Gomez J, Ribeiro ALA, Martinez-Rodriguez A. Effects of Plyometric Jump Training in Sand or Rigid Surface on Jump-Related Biomechanical Variables and Physical Fitness in Female Volleyball Players. Int J Environ Res Public Health. 2021 Dec 11;18(24):13093. doi: 10.3390/ijerph182413093. PMID 34948702
- [Result] Keoliya AA, Ramteke SU, Boob MA, Somaiya KJ. Enhancing Volleyball Athlete Performance: A Comprehensive Review of Training Interventions and Their Impact on Agility, Explosive Power, and Strength. Cureus. 2024 Jan 31;16(1):e53273. doi: 10.7759/cureus.53273. eCollection 2024 Jan. PMID 38435930
- [Result] Mikolajec K, Nowak B, Banys D, Krzysztofik M, Skalski DT, Markiel A, Maszczyk A. Factors determining sports results in elite national volleyball teams between 2004 and 2016. Biol Sport. 2025 Jan;42(1):145-150. doi: 10.5114/biolsport.2025.139085. Epub 2024 Jul 31. PMID 39758186